CLINICAL TRIAL: NCT05508594
Title: Analgesic Efficacy and Pharmacokinetic-pharmacodynamic Relationship of Intranasally Administered Sufentanil, Ketamine, and CT001 After Impacted Mandibular Third Molar Extraction - A Double-blind, Randomised, Placebo-controlled Study
Brief Title: Efficacy and Pharmacokinetic-Pharmacodynamic Relationship of Intranasally Administered Sufentanil, Ketamine, and CT001
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cessatech A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDC 01-0205
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Sufentanil; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- CT001 (Experimental)
  Interventions: Drug: CT001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Sufentanil 27 mcg (Active Comparator)
  Interventions: Drug: Sufentanil
- Ketamine 27 mg (Active Comparator)
  Interventions: Drug: Ketamine
- Sufentanil 13 mcg (Active Comparator)
  Interventions: Drug: Sufentanil
- Ketamine 13 mg (Active Comparator)
  Interventions: Drug: Ketamine
- Sufentanil 40 mcg (Active Comparator)
  Interventions: Drug: Sufentanil
- Ketamine 40 mg (Active Comparator)
  Interventions: Drug: Ketamine
- Sufentanil 13 mcg/Ketamine 13 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 13 mcg/Ketamine 27 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 13 mcg/Ketamine 40 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 27 mcg/Ketamine 13 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 27 mcg/Ketamine 40 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 40 mcg/Ketamine 13 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 40 mcg/Ketamine 27 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine
- Sufentanil 40 mcg/Ketamine 40 mg (Active Comparator)
  Interventions: Drug: Sufentanil; Drug: Ketamine

INTERVENTIONS:
Drug: CT001 — Intranasal
  Arms: CT001
Drug: Placebo — Intranasal
  Arms: Placebo
Drug: Sufentanil — Intranasal
  Arms: Sufentanil 13 mcg; Sufentanil 13 mcg/Ketamine 13 mg; Sufentanil 13 mcg/Ketamine 27 mg; Sufentanil 13 mcg/Ketamine 40 mg; Sufentanil 27 mcg; Sufentanil 27 mcg/Ketamine 13 mg; Sufentanil 27 mcg/Ketamine 40 mg; Sufentanil 40 mcg; Sufentanil 40 mcg/Ketamine 13 mg; Sufentanil 40 mcg/Ketamine 27 mg; Sufentanil 40 mcg/Ketamine 40 mg
Drug: Ketamine — Intranasal
  Arms: Ketamine 13 mg; Ketamine 27 mg; Ketamine 40 mg; Sufentanil 13 mcg/Ketamine 13 mg; Sufentanil 13 mcg/Ketamine 27 mg; Sufentanil 13 mcg/Ketamine 40 mg; Sufentanil 27 mcg/Ketamine 13 mg; Sufentanil 27 mcg/Ketamine 40 mg; Sufentanil 40 mcg/Ketamine 13 mg; Sufentanil 40 mcg/Ketamine 27 mg; Sufentanil 40 mcg/Ketamine 40 mg

SUMMARY:
A randomised, double-blind, parallel-group, study comparing the analgesic effect of intranasal CT001 to intranasal sufentanil, intranasal ketamine or placebo for treatment of acute pain in adults undergoing surgical removal of an impacted mandibular third molar, where bone removal is judged to be needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (The American Society of Anaesthesiologists' Physical Classification System (ASA) I-II) male or female participants scheduled for surgical removal of an impacted mandibular third molar, where bone removal is judged to be needed
* Age: ≥ 18 and < 56 years
* Body Mass index above (>)18.5 or below (<) 30.0 kg/m2
* Prior to randomisation: Numeric Pain Rating Scale (NRS anchored by 0 = "no pain", 10 = "worst pain imaginable") ≥ 5 at rest within 4 hours after the administration of the last dose of local anaesthetic

Exclusion Criteria:

* Current or history of any clinically significant disease or disorder, which, in the opinion of the investigator, may put the potential subject at risk when participating in the study, or influence the potential subject's ability to participate in the study or influence the study results.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of investigational product that is likely to introduce additional risk factors, jeopardize study integrity, or to interfere with the study assessments or procedure
* History of increased bleeding tendency
* Clinically significant mental illness
* Opioid Risk Tool score of >3
* Pain Catastrophizing Scale score, total points >30
* Hospital Anxiety and Depression Scale (HADS), points ≥ 11 for anxiety or ≥ 11 points for depression
* Daily intake of analgesics
* History of alcohol or drug abuse or use of illicit drugs or positive screen for drugs of abuse at screening or on admission to the Clinic prior to the administration of the investigational product.
* Abnormal nasal cavity/airway

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Sum of pain intensity differences at 55 min | 0-55 min
  Derived from pain intensity scores measured by the Numerical Rating Scale (0-10, 0= no pain, 10= worst possible pain).
PK-PD relationship for analgesic efficacy IN sufentanil, IN ketamine and IN CT001 | 0-180 min
  To assess the relationship between analgesic efficacy and the plasma concentrations of intranasal sufentanil, intranasal ketamine and intranasal CT001.

SECONDARY OUTCOMES:
Maximum Pain intensity difference (PIDmax) | 0-180 min
Time to meaningful pain relief | 0-180 min
  Time when participants feel that the pain relief becomes meaningful to them
Sum of pain intensity differences at 30 min | 0-30 min
  Derived from pain intensity scores measured on the Numerical Rating Scale (0-10, 0= no pain, 10= worst possible
Rescue medication | 0-180 min
  Number of participants receiving rescue medication
Number of patients who are considered a responder/non-responder, 30% | 0-30 min
  Number of participants with at least 30% reduction in pain intensity score compared to baseline
Number of patients who are considered a responder/non-responder, 50% | 0-30 min
  Participants with at least at least 50% reduction in pain intensity score compared to baseline
Sum of pain intensity differences at 90 min | 0-90 min
  Derived from pain intensity scores measured on the Numerical Rating Scale (0-10, 0= no pain, 10= worst possible
Time to perceptible pain relief | 0-180 min
  Time when participants feel that the pain relief becomes meaningful to them
Time to rescue medication | 0-180 min
Mean pain intensity difference (PID) from baseline at rest | 0-180 min
Mean pain intensity difference (PID) from baseline on jaw movement | 0-181 min
Ramsay sedation score | 0-179 min
  Change from baseline in Ramsay sedation score (1= agitated, anxious, restless, 6= unarousable)
Median time to a request for rescue medication | 0-180 min

CONTACTS AND LOCATIONS:
Locations (1):
- DanTrials, Copenhagen, NV, Denmark